CLINICAL TRIAL: NCT05025761
Title: A Personal Protection Package for Reducing Malaria Transmission in Forest-going Mobile and Migrant Populations in Myanmar: A Stepped-wedge Trial With Nested Mixed-methods Study
Brief Title: Reducing Malaria Transmission in Forest-going Mobile and Migrant Populations in Myanmar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Macfarlane Burnet Institute for Medical Research and Public Health Ltd (Other)
Collaborators: Health Poverty Action (Other); National Malaria Control Program, Myanmar (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 260/21_forest_Myanmar
Record Dates: First submitted 2021-08-16; First posted 2021-08-27 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-08

CONDITIONS: Plasmodium Falciparum Infection
Keywords: malaria; prevention; vector; migrant; elimination; vivax; falciparum; community-delivered; intervention
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster-randomized controlled trial (one-way crossover) with nested mixed methods study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personal protection package (Experimental): A personal protection package that includes Long-lasting insecticidal hammock net (LLIHN),insect repellent (DEET), Insecticide-treated clothes (ITC), and mobile and migrant population-tailored behavioural change communication (BCC) package
  Interventions: Other: Personal protection package
- Control (No Intervention): No personal protection package

INTERVENTIONS:
Other: Personal protection package — The personal protection package will be distributed to mobile and migrant peoples in each village according to the stepped wedge design.
  Arms: Personal protection package

SUMMARY:
This stepped-wedge cluster-randomized controlled trial with nested mixed methods study will assess the effectiveness, acceptability, feasibility and cost effectiveness of a personal protection package to reduce malaria transmission among mobile and migrant populations (MMPs) and the general population in their residing villages in Myanmar.

DETAILED DESCRIPTION:
Over the last decade, the burden of malaria has fallen dramatically in the Greater Mekong Subregion, with deaths falling by 95% and cases by 76% between 2012 and 2019.The declining malaria burden in GMS has largely been attributed to the deployment of interventions of malaria prevention tools such as long-lasting Insecticidal Nets (LLIN), and widespread availability of rapid diagnostic tests and artemisinin combination therapies. However, residual transmission exists among high risk populations, particularly mobile and migrant populations who enter forests for work. New interventions targetting these high risk groups are needed if countries of the Greater Mekong Subregion are to achieve malaria elimination by 2030. The study will be conducted in malaria endemic areas of Myanmar which have large forest going MMP populations. The aim of the study is to assess the effectiveness, acceptability, feasibility and cost-effectiveness of a personal protection package to reduce malaria transmission among mobile and migrant populations (MMPs) and the general population in their residing villages in Myanmar. The personal protection package includes WHO prequalified long-lasting insecticidal net (LLIN), insect repellent (N, N-Diethyl-meta-toluamide (DEET), insecticide-treated clothes (ITC), and a MMP-tailored behavioural change communication (BCC) package. The study design is a stepped-wedge cluster-randomized controlled trial with nested mixed methods study. The stepped-wedge cluster randomized trial will estimate the effectiveness of a personal protection package provided to forest-going MMPs (the intervention) delivered by village malaria volunteers at the site (village/worksite) level on reducing Plasmodium spp. infections (primary outcome). Whilst the personal protection package will be provided to mobile and migrant populations in each village in a step-wise manner, primary and secondary outcomes relating to malaria testing will be collected in all consenting individuals in the village who present for malaria rapid diagnostic tests, whether they are mobile and migrant people or not. The study will also include investigation of antibody responses to Plasmodium spp. and mosquito vectors and molecular markers of antimalarial drug resistance.

The study will be implemented between July 2021 (M1) to June 2022 (M12). The personal protection package for MMPs will be implemented sequentially in a minimum of 100 villages serviced by an ICMV. The villages will be grouped into 11 blocks of 9 villages, with each block transitioned from control phase (before introduction of the personal protection package) to intervention phase (after introduction of the personal protection package) at monthly intervals in random order. This follows an initial one-month baseline period at the start of the study period where all villages will not be exposed to the personal protection package exclusively.

For this proposed stepped-wedge cluster randomized controlled study, it is estimated that approximately 30 RDTs per month will be tested in each study site (village/worksite) and there will be 36,000 MMP tests over 12 months in 100 villages/worksites. It will be undertaken yielding a relative minimum detectable difference of 40% in odds of RDT-detectable malaria infection (assuming a village intraclass correlation [ICC]= 0.42 [6]; 5% significance; 80% power and 1% RDT malaria prevalence).

For the stepped-wedged cluster randomized trial, both descriptive and primary outcome trial analyses will be performed. In both analyses, sampling weights will be derived and applied in analyses where village selection probabilities are not equal - possible if the achieved number of villages sampled across townships varies. Furthermore, cluster robust standard errors will be used in all descriptive analyses given the complex sampling design. Differences in prevalence of malaria infections will be estimated across intervention and control periods using generalized linear mixed modelling (e.g. logit link function and binomial distribution).

ELIGIBILITY:
Inclusion Criteria for states/regions:

* Capacity of Burnet Institute Myanmar to conduct field implementation
* Presence of ICMV networks managed by NMCP and HPA
* High malaria burden
* High MMP activities
* Available budget

Exclusion Criteria for states/regions:

* The township does not have an NMCP or HPA-provided ICMV network
* The township is not under the administration of NMCP or HPA
* The township has an ongoing armed conflict at the time of sampling
* The location of the township is not geographically or politically feasible for the NMCP or HPA staff to conduct regular supervision visits

Exclusion criteria for villages:

* The village has no malaria cases or API less than 1 in any of the past three years (2018 - 2020)
* The village has no MMPs
* The village has no ICMVs actively working in the village
* The village has a government health facility for malaria services
* The village has an ICMV program operated by any organizations other than NMCP or HPA

Inclusion Criteria for MMP participants (personal protection package intervention):

* Currently living in the selected villages/ worksites
* Being any of the following types of workers: Traditional slash-and-burn and paddy field farming communities visiting their forest farms (commonly ethnic minority groups); Seasonal agricultural laborers; Forest workers in the informal sector (hunters, small-scale gem/gold miners, people gathering forest products (precious timber, construction timber, rattan/bamboo); Transient or mobile camp residents associated with commercial projects (road/pipeline construction, large-scale logging, deep seaport projects, etc.); Formal and informal cross-border migrant workers
* Aged 18 years and over

Inclusion criteria for the focus group discussion:

• Participants selected purposively from the same cohort of MMPs who have received the personal protection package during the study period

Inclusion criteria for semi-structured interviews with local health stakeholders:

* Aged over 18 years
* From different levels of NMCP, EHOs and HPA
* Basic health staff such as Public Health Supervisors, Midwives, Health Assistants, Township Health Officers and focal person from Township VBDC/NMCP offices
* Health staff from ethnic health organizations such as medics, doctors and nurses
* Health staff from HPA such as field supervisor, field office manager, technical officer

Inclusion criteria for semi-structured interviews with ICMVs:

• ICMV participants will be selected purposively from the ICMVs actively working in the selected villages.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Plasmodium spp. infection diagnosed by RDT | Assessed weekly, longitudinally over 12 months
  Change in the number of Plasmodium spp. infections detected by RDT per week per village (SD Bioline P.f/P.v)

SECONDARY OUTCOMES:
Symptomatic malaria diagnosed by RDT | Assessed weekly, longitudinally over 12 months
  Change in the number of symptomatic Plasmodium spp. infections detected by RDT per week per village
Plasmodium spp. infection as determined by polymerase chain reaction (PCR) | Assessed weekly, longitudinally over 12 months
  Change in the number of Plasmodium spp. infections as determined by PCR using from RDT cassettes and dried blood spots
Plasmodium spp. drug resistance mutations | Assessed weekly, longitudinally over 12 months
  Prevalence and change in the number of Plasmodium spp. drug resistance mutations as determined by PCR from RDT cassettes and dried blood spots
Prevalence of antibodies to Plasmodium spp. | Assessed weekly, longitudinally over 12 months
  Prevalence of antibodies to Plasmodium spp. determined by Enzyme Linked Immunosorbent assay (ELISA) from RDT and DBS samples
Levels of antibodies to Plasmodium spp. | Assessed weekly, longitudinally over 12 months
  Levels of antibodies to Plasmodium spp. determined by Enzyme Linked Immunosorbent assay (ELISA) from RDT and DBS samples
Prevalence of antibodies to vector salivary antigens | Assessed weekly, longitudinally over 12 months
  Prevalence of antibody biomarkers of vector exposure determined by Enzyme Linked Immunosorbent assay (ELISA) from RDT and DBS samples
Levels of antibodies to vector salivary antigens | Assessed weekly, longitudinally over 12 months
  Levels of antibody biomarkers of vector exposure determined by Enzyme Linked Immunosorbent assay (ELISA) from RDT and DBS samples
Levels of knowledge, attitude and practice regarding malaria prevention among MMPs (qualitative research) | At 12 months
  Focus group discussions
Proportion of survey respondents (MMPs) who accept and are willing to use/ did use the personal protection package according to the protocol | At 12 months
  Focus group discussions; Questionnaire

IPD SHARING:
Plan to Share IPD: No